CLINICAL TRIAL: NCT03053245
Title: Mobile Critical Care Recovery Program for Acute Respiratory Failure Survivors
Acronym: m-CCRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Babar Khan, MD, MS, Assistant Professor of Medicine Research Scientist, Regenstrief Institute, Inc. Research Scientist, Indiana University Center for Aging Research, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01HL131730 (NIH)
Record Dates: First submitted 2017-02-01; First posted 2017-02-15 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Acute Respiratory Failure; Post-Intensive Care Syndrome
Keywords: Collaborative Care Model; Intensive Care Unit
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Critical Care Recovery Program (Experimental): The group will receive the Mobile Critical Care Recovery Program (m-CCRP) intervention which includes care coordination and collaborative care model for one year post enrollment.
  Interventions: Behavioral: Mobile Critical Care Program
- Attention Control (Active Comparator): The attention control group will receive telephone based check ins related to their health from the research study team.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Mobile Critical Care Program — The m-CCRP revolves around the central figure of a care coordinator who will organize and align recovery resources. The care coordinator is a registered nurse whose scope of practice includes health coaching, case managing, community organizing, and nursing care provider. The m-CCRP support team will consist of a critical care physician (Dr. Khan), a geriatrician with expertise in collaborative care (Dr. Boustani), an ICU collaborative care nurse (Dr. Lasiter), and a psychologist (Dr. Unverzagt). This team will meet weekly with the care coordinator. Drs. Khan and Boustani will be accessible to the coordinator through phone or pager at all times.
  Arms: Mobile Critical Care Recovery Program
Behavioral: Attention Control — Patients in this group will receive regular wellness calls from the research team.
  Arms: Attention Control

SUMMARY:
The m-CCRP randomized controlled trial will evaluate the efficacy of a collaborative critical care recovery program from acute respiratory failure (ARF) survivors in accomplishing the Institute of Healthcare Improvement's triple aims of better health, better care, at lower cost.

Primary Aim:

To assess the efficacy of m-CCRP in improving the QOL of ARF survivors compared to attention control at twelve months post hospital discharge.

Secondary Aims:

1. To evaluate the efficacy of m-CCRP in improving cognitive, physical, and psychological function of ARF survivors at twelve months post hospital discharge when compared to attention control.
2. To evaluate the efficacy of m-CCRP in reducing health-care utilization, defined as time from enrollment to emergency department visits and/or hospital re-admission, by ARF survivors as compared to attention control at twelve months post hospital discharge.

DETAILED DESCRIPTION:
Five million Americans require admission to intensive care units (ICU) annually due to life threatening illnesses, and this number is expected to rise.4 Two million of these ICU admissions are secondary to Acute Respiratory Failure (ARF) with more than half requiring mechanical ventilation. Greater than 50% of the patients with ARF who survive their ICU stay suffer from long-term morbidity in the form of functional disability, cognitive disability, major or minor depression, and anxiety. These complications negatively impact the quality of life (QOL) of ARF survivors, interfere with their physical and emotional recovery, and lead to long-term disability with less than half of ARF survivors returning to the work force. Ongoing care for ARF survivors has been estimated to cost $3.5 million per ARF survivor at 1 year. This constellation of ICU sequelae with attendant morbidity has been designated as the post-intensive care syndrome (PICS). There are community resources and rehabilitation services available to ARF survivors, but the current fragmented nature of our healthcare system is unable to integrate and coordinate care in order to provide the most meaningful recovery.

The Institute of Medicine recommends the development of care coordination programs to deliver patient-centered and interdisciplinary-based medical care. Indiana University Center for Aging Research (IUCAR) has over 20 years of experience in delivering interdisciplinary, collaborative care through pragmatic interventions utilizing care coordinators. Care coordinator delivery models have improved care of patients with dementia, depression, functional decline and PICS. Our PICS clinic, the Critical Care Recovery Center (CCRC) was developed in 2011 to enhance cognitive, physical, and psychological recovery of ICU survivors.

Since then, CCRC has provided care to over 200 survivors with a high burden of PICS (88% had cognitive impairment; 60% had depression). CCRC showed feasibility and initial efficacy in managing PICS. However given its traditional outpatient clinic structure, CCRC has limited physical access to ARF survivors, leading to delayed evaluation and an added travel burden on ARF survivors. Building from the experience of the CCRC and our other successful care coordinator based programs; we now propose a mobile model of post-ICU collaborative care with greater access to enhance the recovery of ARF survivors.

The overarching aim of the proposed program is to improve the QOL of patients who survived an episode of ARF by maximizing their cognitive, physical, and psychological recovery utilizing a mobile care coordinator. The care coordinator will bring the intervention to the patient irrespective of the patient's physical location and will be supported by an interdisciplinary team of a critical care physician, a health services scientist, an ICU nurse, and a psychologist, with input from other consultants as needed. In addition, dynamic feedback through process measurement tools and care coordination support software will inform the recovery process. We propose to evaluate the efficacy of our collaborative care intervention termed the "Mobile Critical Care Recovery Program (m-CCRP)" through a randomized clinical trial among survivors of ARF.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Hospitalized in the ICU
* Diagnosed with Acute Respiratory Failure (ARF) requiring greater than or equal to 24 hours of mechanical ventilation or noninvasive positive pressure ventilation or high flow nasal canula.
* Discharged to home, skilled nursing facility, sub-acute rehabilitation care, or long-term acute care
* English speaking
* Able to consent either in-person or through legally authorized representative
* Have access to a telephone

Exclusion Criteria:

* Hospitalized to a regular non-ICU ward
* Diagnosis of cancer with life expectancy less than 1 year
* Admitted with ischemic or hemorrhagic cerebrovascular accident, traumatic brain injury, or undergoing neurosurgery
* History of dementing illnesses and other neurodegenerative disease such as Alzheimer's disease, Parkinson's disease, or vascular dementia
* Unable to complete study questionnaire due to severe hearing loss
* Legally blind
* Pregnant (assessed by urine pregnancy test) or nursing
* Living outside the greater Indianapolis area
* Recent history of alcohol or substance abuse
* Status post tracheostomy and not eligible for a speaking valve
* Incarcerated at the time of study enrollment
* Schizophrenia or bipolar disorder (confirmed by EMR)
* Homelessness
* Illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Babar A Khan, MD, MS, Principal Investigator — Indiana University Center for Aging Research
Locations (3):
- United States (3):
  - Eskenazi Hospital, Indianapolis, Indiana
  - Methodist Hospital, Indianapolis, Indiana
  - University Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Savsani PK, Khan SH, Perkins AJ, Wang S, Jawaid S, Moiz S, Monahan PO, Kroenke K, Gao S, Khan BA. Performance of the Healthy Aging Brain Care Monitor Self Report in Monitoring Post-Intensive Care Syndrome Among Acute Respiratory Failure Survivors. Crit Care Med. 2025 Feb 1;53(2):e341-e352. doi: 10.1097/CCM.0000000000006522. Epub 2024 Nov 11. PMID 39526840
- [Derived] Khan BA, Perkins AJ, Khan SH, Unverzagt FW, Lasiter S, Gao S, Wang S, Zarzaur BL, Rahman O, Eltarras A, Qureshi H, Boustani MA. Mobile Critical Care Recovery Program for Survivors of Acute Respiratory Failure: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2353158. doi: 10.1001/jamanetworkopen.2023.53158. PMID 38289602
- [Derived] Khan S, Biju A, Wang S, Gao S, Irfan O, Harrawood A, Martinez S, Brewer E, Perkins A, Unverzagt FW, Lasiter S, Zarzaur B, Rahman O, Boustani M, Khan B. Mobile critical care recovery program (m-CCRP) for acute respiratory failure survivors: study protocol for a randomized controlled trial. Trials. 2018 Feb 7;19(1):94. doi: 10.1186/s13063-018-2449-2. PMID 29415760

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol subjects were considered to be enrolled in the study at the time of completion of the informed consent process. 503 subjects were enrolled. 466 subjects were randomized to one of the two study groups.
Period: Overall Study
Arm/Group | Mobile Critical Care Recovery Program | Attention Control
Started | 233 | 233
Completed | 153 | 147
Not Completed | 80 | 86

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Critical Care Recovery Program | Attention Control | Total
Number analyzed (Participants) | 233 | 233 | 466
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (14.3) | 56.9 (14.4) | 56.1 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 125 | 250
  Male | 108 | 108 | 216
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  Not Hispanic or Latino | 233 | 228 | 461
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 94 | 78 | 172
  White | 134 | 146 | 280
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Self Reported Quality of Life PCS: Physical Component Score at 1 Year
Description: Utilizing SF-36 The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) consists of eight domains. It yields two summary scores (PCS: physical component score, and MCS: mental component score). MCS and PCS range from 0 to 100, and higher scores indicate better health status. A difference of 2 or more points is considered clinically meaningful for both the PCS and MCS subscales of SF-36.
Time Frame: 1 year
Population: Only participants who were able to complete the scale are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Critical Care Recovery Program | Attention Control
Number analyzed (Participants) | 153 | 146
score on a scale | 36.22 (12.55) | 35.29 (12.20)

2. Primary Outcome: Self Reported Quality of Life MCS: Mental Component Score at 1 Year
Description: as for outcome 1
Time Frame: 1 year
Population: Only participants who were able to complete the scale are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Critical Care Recovery Program | Attention Control
Number analyzed (Participants) | 153 | 146
score on a scale | 49.81 (11.75) | 51.12 (10.23)

3. Primary Outcome: Cognitive Assessment Score at 1 Year
Description: Utilizing RBANS: Repeatable Battery for the Assessment of Neuropsychological Status.
  The overall RBANS z-score is the mean of the 7-item (RBANS subscale) z-scores that could be collected in person and by phone. The 7 subscales are: List Learning, Story Memory, Semantic fluency, Digit Span, List Recall, List Recognition, Story Recall.
  A Z-Score of 0 is the population mean. Values above 0 represent better outcomes.
Time Frame: 1 year
Population: Only participants who were able to complete the scale are included in the analysis.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Mobile Critical Care Recovery Program | Attention Control
Number analyzed (Participants) | 129 | 133
Z-score | 0.27 (0.70) | 0.26 (0.68)

4. Secondary Outcome: Depression Symptoms at 1 Year
Description: PHQ-9 (Patient Health Questionnaire-9) Scores range from 0 to 27 on the PHQ-9 with higher scores indicating greater severity of depression.
Time Frame: 1 year
Population: Only participants who were able to complete the scale are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Critical Care Recovery Program | Attention Control
Number analyzed (Participants) | 153 | 147
score on a scale | 5.94 (6.13) | 5.66 (5.37)

5. Secondary Outcome: Anxiety Symptoms at 1 Year
Description: GAD-7 (Generalized Anxiety Disorder-7) Scores range from 0 to 21 on the GAD-7 with higher scores greater anxiety.
Time Frame: 1 year
Population: Only participants who were able to complete the scale are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Critical Care Recovery Program | Attention Control
Number analyzed (Participants) | 153 | 147
score on a scale | 5.04 (6.08) | 4.82 (5.25)

6. Secondary Outcome: Physical Performance at 1 Year
Description: Utilizing SPPB The Short Physical Performance Battery (SPPB) will measure physical training effects on balance and strength.
  Ranges from 0-12: higher score is better outcome
Time Frame: 1 year
Population: Only participants who were able to complete the scale are included in the analysis. Post COVID-19 no SPPB Tests were performed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Critical Care Recovery Program | Attention Control
Number analyzed (Participants) | 34 | 32
score on a scale | 8.8 (3.0) | 8.7 (2.8)

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events from the time of informed consent process completion until the end of study participation. This was approximately 1 year if the study was completed.
Arm/Group | Mobile Critical Care Recovery Program | Attention Control
All-Cause Mortality (participants affected / at risk) | 24/233 | 38/233
Serious Adverse Events (participants affected / at risk) | 0/233 | 0/233
Other Adverse Events (participants affected / at risk) | 0/233 | 0/233

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/45/NCT03053245/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/45/NCT03053245/ICF_001.pdf